CLINICAL TRIAL: NCT00473148
Title: Weaning of Mechanical Ventilation Guided by the Natriuretic Peptide of Type B
Brief Title: B-type Natriuretic Peptide for the Management of Weaning
Acronym: BMW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Dräger Médical S.A (Unknown); Abbott RDx Cardiometabolic (Other)
Responsible Party: Christophe AUCAN: Manager, Department of Clinical Research and Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P051018
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2008-11

CONDITIONS: Respiratory Insufficiency
Keywords: Duration of weaning from invasive ventilation; Mechanical ventilation; Weaning; B-type natriuretic peptide; Fluid balance; Diuretics; Intubated patient receiving mechanical ventilation; for at least 24 hours; Respiratory insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): BNP-guided treatment (Furosemide)
  Interventions: Procedure: BNP-guided weaning
- 2 (No Intervention)
  Interventions: Procedure: Standard physician-directed weaning

INTERVENTIONS:
Procedure: BNP-guided weaning — BNP-guided weaning
  Arms: 1
Procedure: Standard physician-directed weaning — Standard physician-directed weaning
  Arms: 2

SUMMARY:
Several clinical findings and clinical trials have suggested that the prognosis of intensive care unit (ICU) patients may be improved by minimizing the positive fluid balance. In particular, a global vascular overload could lead to weaning failure. The purpose of this international, multicenter, controlled, randomized trial is to test if the incorporation of a B-type natriuretic peptide (BNP) assay in a mechanical ventilation weaning protocol helps optimize the weaning process and reduce the duration of the ventilatory weaning period.

DETAILED DESCRIPTION:
Mechanical ventilation may give rise to complications with an incidence that increases with the duration of respiratory support. The purpose of the weaning procedure is to reduce the duration of mechanical ventilation without incurring a substantial risk of failure. Several clinical findings and clinical trials have suggested that the prognosis of ICU patients may be improved by minimizing the positive fluid balance. In particular, a global vascular overload could lead to weaning failure. B-type natriuretic peptide (BNP) is a hormone secreted by the ventricular cardiomyocytes in response to increased wall stretch, and its plasma levels are correlated with left ventricular filling pressure. In a preliminary study on 102 patients undergoing weaning from mechanical ventilation, the baseline BNP levels before weaning were found to be an independent risk factor for weaning failure. In surviving patients, BNP levels were significantly correlated with the duration of weaning procedure. The purpose of this international, multicenter, controlled, randomized trial is to test if the incorporation of a BNP assay in a mechanical ventilation weaning protocol helps optimize the weaning process and reduce the duration of ventilatory weaning period. Patients on mechanical ventilation presenting weaning criteria will be randomly assigned to two groups (standard physician-directed weaning or weaning guided by BNP assay). In order to standardize the weaning process, patients will be ventilated with an automatic computer-driven weaning system in the two groups (EVITA Smart Care System, Drager Medical). A blood sample will be collected from all patients every morning for BNP assay by the rapid immunofluorescence test (Triage BNP Test, BIOSITE). In the control group, the clinician will not be informed about the assay results and weaning will be carried out according to usual practices. Patients in the intervention group will receive diuretics according to a clinical practice algorithm based on plasma BNP levels and a fluid intake restriction. The primary endpoint for the two groups will be duration of weaning from mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Intubated patient receiving mechanical ventilation for at least 24 hours
* SpO2 ≥ 90% with FiO2 ≤ 50% and PEP ≤ 8 cm H2O
* Hemodynamic stability without vasopressor therapy (dopamine ≤ 10 γ/kg/min and dobutamine ≤ 10 γ/kg/min are however allowed) nor fluid bolus (rapid infusion of at least 500 ml of macromolecules or 1000 ml of saline) during the twelve previous hours
* Sedation stopped or reduced during the previous 48 hours (analgesia may be continued)
* Stable neurological status with Ramsay score ≤ 5
* Body temperature > 36.0 °C and < 39 °C
* Informed consent signed by patient or close relative

Exclusion Criteria:

I: Definite exclusion criteria:

* Pregnancy or lactation
* Age < 18 years
* Known allergy to furosemide or sulphonamides
* Tracheotomy on inclusion
* Hepatic encephalopathy
* Cerebral edema, acute hydrocephaly
* Myasthenia gravis or acute idiopathic polyradiculoneuritis (Guillain-Barré syndrome)
* Decision to withdraw life support
* Prolonged cardiac arrest with poor neurological prognosis

II: Temporary exclusion criteria:

* Extubation of the patient programmed for the same day
* Acute right ventricular insufficiency (pulmonary embolism, right myocardial infarction)
* Renal insufficiency defined by one of the following: renal replacement therapy, or plasma urea > 25 mmol/L, or plasma creatinine > 180 µmol/L, or creatinine clearance < 30 mL/min or increase by more than 25% of plasma creatinine during the previous 24 hours
* One of the following metabolic abnormalities: blood sodium > 150 mEq/L; blood potassium < 3.5 mEq/L; metabolic alkalosis with arterial pH > 7.50
* Injection of iodinated contrast agent during the preceding six hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Duration of weaning from invasive ventilation | during ventilation

SECONDARY OUTCOMES:
Total duration of weaning from invasive and noninvasive ventilation | during hospitalisation
Total duration of mechanical ventilation | during hospitalisation
Length of stay in the ICU, length of stay in hospital, number of complications in intensive care, number of prolonged weanings (> 15 days), number of cases of nosocomial pneumonia, number of successful extubations, extubation complication rates | during hospitalisation in ICU
Cost of stay in the ICU | in the ICU
Cost of stay in hospital | during the all stay
Mortality in ICU | in ICU
Mortality sixty days after randomization | sixty days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Armand Mekonto Dessap, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CHU Henri Mondor, Créteil, France

REFERENCES:
- [Derived] Dessap AM, Roche-Campo F, Launay JM, Charles-Nelson A, Katsahian S, Brun-Buisson C, Brochard L. Delirium and Circadian Rhythm of Melatonin During Weaning From Mechanical Ventilation: An Ancillary Study of a Weaning Trial. Chest. 2015 Nov;148(5):1231-1241. doi: 10.1378/chest.15-0525. PMID 26158245
- [Derived] Mekontso Dessap A, Katsahian S, Roche-Campo F, Varet H, Kouatchet A, Tomicic V, Beduneau G, Sonneville R, Jaber S, Darmon M, Castanares-Zapatero D, Brochard L, Brun-Buisson C. Ventilator-associated pneumonia during weaning from mechanical ventilation: role of fluid management. Chest. 2014 Jul;146(1):58-65. doi: 10.1378/chest.13-2564. PMID 24652410
- [Derived] Mekontso Dessap A, Roche-Campo F, Kouatchet A, Tomicic V, Beduneau G, Sonneville R, Cabello B, Jaber S, Azoulay E, Castanares-Zapatero D, Devaquet J, Lellouche F, Katsahian S, Brochard L. Natriuretic peptide-driven fluid management during ventilator weaning: a randomized controlled trial. Am J Respir Crit Care Med. 2012 Dec 15;186(12):1256-63. doi: 10.1164/rccm.201205-0939OC. Epub 2012 Sep 20. PMID 22997204